CLINICAL TRIAL: NCT03302858
Title: A Safety and Efficacy Trial of Circumferential Anal Canal Radiofrequency Ablation for High-Grade Anal Intraepithelial Neoplasia Using the BARRX™ Anorectal Wand
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stephen E. Goldstone (Other)
Responsible Party: Sponsor-Investigator, Stephen E. Goldstone, Surgeon, Laser Surgery Care
Organization: Laser Surgery Care (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-2017
Record Dates: First submitted 2017-09-20; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: HSIL, High Grade Squamous Intraepithelial Lesions; Anal Cancer; HPV-Related Squamous Cell Carcinoma; Human Papilloma Virus; Human Papillomavirus Infection; Ain III
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Anus Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: BARRX™ Anorectal Wand — The radiofrequency ablation (RFA) or Barrx™ Ablation System used in this protocol comprises an RFA generator (Barrx™ FLEX) and the Barrx™ Anorectal Wand. The generator and wand are cleared by the FDA for human use and the wand is specifically cleared for treatment of anal neoplasia. The present FDA indication for use statement is: "The Barrx™ catheters are indicated for use in the coagulation of bleeding and non-bleeding sites in the gastrointestinal tract including, but not limited to, the esophagus. Indications include esophageal ulcers, Mallory-Weiss tears, arteriovenous malformations, angiomata, Barrett's esophagus, Dieulafoy lesions, angiodysplasia, gastric antral vascular ectasia, and radiation proctitis."

SUMMARY:
The purpose of this research is to assess the safety and effectiveness of circumferential radiofrequency ablation (RFA) to the anal canal using the BarrxTM Ablation System to destroy anal high-grade squamous intraepithelial lesions (HSIL). The BarrxTM Ablation System used in this study comprises an RFA generator (Barrx™ FLEX) and the BarrxTM Anorectal Wand. The generator and wand are cleared by the Food and Drug Administration (FDA) for human use and the wand is specifically cleared for treatment of anal intraepithelial neoplasia (AIN). AIN is a precancerous condition. HSIL is an advanced form of AIN. The presence of HSIL has traditionally warranted treatment. RFA has been shown in many studies to effectively and safely destroy precancerous cells in a condition called Barrett's esophagus, which is a precancerous condition of the esophagus (the swallowing tube). Recent studies have shown that RFA may offer the same benefits for those with HSIL in the anal canal. In particular, ablation of the entire circumference of the canal seems to reduce recurrence of HSIL in other locations of the anal canal.

This study will last between 12 to 15 months. Subjects will be required to undergo 5 to 8 study visits as outlined below that are carried out by the study doctors or the physician assistant. Most visits will last approximately one hour. Some may be shorter and some may be longer. Up to seventy (70) volunteers will participate in this study at several locations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. HRA 2 to 8 weeks prior to the 0 month RFA visit yielding one or more flat, non- condylomatous biopsy-proven HSILs that are

   * Located entirely within the eligible treatment zone AND
   * Contiguous with the squamocolumnar junction
3. Eligible treatment zone (ETZ) is defined as

   * 3 cm above the dentate line to the anocutaneous line AND
   * Full anorectal circumference
4. If female of child-bearing age, negative pregnancy test within 8 weeks of the 0 month RFA visit and declared intent to remain on birth control throughout the trial, or declaration of infertility defined as subject report of status as post-menopausal or surgically sterile (status post hysterectomy or tubal ligation).
5. If HIV positive

   * HIV positive on antiretroviral therapy for at least 3 months with laboratory blood work within 12 weeks prior to the 0 month visit demonstrating viral load < 50
   * CD4 count ≥ 250/mm3
   * ANC > 750/mm3
   * Platelet count ≥ 75,000/mm3
   * Hemoglobin ≥ 9.0 g/dl

Exclusion Criteria:

1. Any biopsy-proven HSIL partially outside of the ETZ (for example, an HSIL lesion with extension to the perianal skin)
2. Any condylomas in the eligible treatment zone > 1/2 cm diameter
3. Any anal or rectal pathology requiring treatment including ulcer, fistula, fissure, or proctitis
4. Any anal stricture or stenosis in patient history or upon examination.
5. Symptomatic scarring in anal canal (i.e. not pliable, hyperkeratosis)
6. History of or present anal or rectal cancer
7. History of pelvic radiation therapy
8. History of HPV vaccination or plans to initiate HPV vaccination during the trial
9. History of ablation or resection therapy within the ETZ within 3 months prior to the 0 month RFA visit (other than cauterization or excision of condylomata)
10. History of topical therapy (e.g. Imiquimod, 5-FU, Trichloroacetic acid) within the

    ETZ within 3 months prior to the 0 month RFA visit
11. Hemorrhoids > grade III
12. Fecal incontinence
13. Concurrent disease requiring systemic immunosuppression therapy
14. Concurrent malignancy requiring systemic therapy
15. Life expectancy < 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Percent of patients who have histologically cleared high-grade squamous intraepithelial lesions (HSIL) at the SCJ at 12 months as measured by HRA | 12 months
  Histologic clearance of all HSIL within the ETZ on a patient and lesion basis at 12 months from first RFA

SECONDARY OUTCOMES:
Persistence of treated HSIL index lesions | 3 months post RFA
Safety of circumferential ablation of anal canal HSIL using the Barrx™ Anorectal Wand as defined by number of patients with adverse events (including prolonged pain, bleeding, anal strictures, etc). | 12 months
Percent of patients who have histologically cleared low-grade squamous intraepithelial lesions (LSIL) at the SCJ at 12 months as measured by HRA | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Laser Surgery Care, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT03302858/Prot_SAP_000.pdf